Approval Date: 1/30/2019



TITLE: Use of Platelet Rich Plasma after Arthroscopic Debridement for Triangular

Fibrocartilage Complex Tears

**SPONSOR:** CEDARS-SINAI MEDICAL CENTER

PARTICIPATING RESEARCHERS: DAVID KULBER, M.D.

PRINCIPAL INVESTIGATOR

STUDY CONTACT PHONE NUMBER AT CSMC: 310-423-5900

**AFTER HOURS CONTACT (24 HOURS): 310-423-5900** 

# 1. WHAT IS THE PURPOSE OF THIS RESEARCH STUDY?

We are doing this study to determine if treatment with platelet rich plasma improves outcomes after arthroscopic debridement for patients with triangular fibrocartilage complex (TFCC) tears. The TFCC is a structure made of cartilage that stabilizes and cushions the bones in the wrist. Injury to the TFCC can cause wrist pain and loss of strength in the hand. Surgical treatment is performed using wrist arthroscopy to clean up damaged structures, which is called debridement. We want to know if there's a difference after arthroscopic debridement in post-operative pain, wrist function and patient satisfaction between those treated with platelet rich plasma and those that are not.

You are being asked to take part in this research study because you have a triangular fibrocartilage complex tear and are a candidate for surgical treatment. The study will enroll up to 48 people in total.

This research study is designed to test the use of platelet-rich plasma (PRP) after arthroscopic debridement.

Plasma is the liquid part of blood that contains blood cells and platelets. Platelets are best known for their role in normal clot formation, but they also contain growth factors that react within the body to initiate healing. Platelet-rich plasma (PRP) is created using a small sample (approximately 9 cc) of the patient's own venous blood, obtained through the patient's IV. The blood is placed in a tube and spun in a machine for 6 minutes, which removes the red and white blood cells from the plasma. The sample is then transferred to a second tube and spun for 15 minutes. What results is plasma with a high concentration of platelets that may be injected into areas of injury to stimulate the natural healing process and reduce inflammation.

Approval Date: 1/30/2019

The PRP will be prepared using the CASCADE Autologous Platelet System. This system has been cleared for marketing, sale and use by the U.S. Food and Drug Administration (FDA) and includes the tubes and solutions used for preparation of the PRP as described above.

PRP has been used in many fields of medicine including orthopedic and plastic surgery to promote healing of soft tissues, tendons, ligaments, and cartilage. It has been used to treat both short and long-term musculoskeletal injuries.

# 2. WHAT WILL HAPPEN DURING THE STUDY?

This section provides a general overview of what will happen during your participation in this study. Information included below should be considered along with the flowchart of procedures attached as Appendix A.

The flowchart shows a timeline for research-related or standard of care procedures that are involved in your participation in this study. **Research-related procedures** are those performed solely for the research. They would not be performed if you did not take part in the study. **Standard of care (routine)** procedures would be performed both as part of this study and if you do not participate in this study.

A table describing procedures done solely for the purposes of monitoring and assessing your condition during this study is attached as Appendix B to the end of this consent form. Standard of care procedures that will be repeated or done at greater frequency are listed in the flow chart, attached Appendix A.

#### Overview of study:

This is a randomized, single-blind research study.

- "Randomized" means that you will be assigned to a study group by chance, like flipping a coin. You will be randomized into one of 2 study groups, and will have an equal chance of being placed in one of the groups described below.
- "Single-blind" means that the researchers will know which group you are assigned to but will not tell you which group you are participating in.

This study has 2 study groups:

- Group A will get the usual arthroscopic debridement for treatment of a triangular fibrocartilage complex tear followed by placebo (normal saline) injection
- Group B will get the usual arthroscopic debridement for treatment of a triangular fibrocartilage complex tear followed by treatment with platelet rich plasma (PRP)

A computer will randomly assign you to a study group. This is done because no one knows if the results experienced by the participants in one study group are better, the same, or worse than the results experienced by participants in the other. Once you are put in one group, you cannot switch to another group. Neither you nor your doctor can choose the group in which you will be placed.

Approval Date: 1/30/2019

Either of these approaches could help your condition but could also cause side effects. This study will allow the researchers to learn whether the different approaches are better, the same, or worse than the current standard of care. Arthroscopic debridement has already been tested for safety and is currently the standard of care. Platelet rich plasma has also been tested for safety; however, it is not currently part of the standard of care.

This is a placebo-controlled study. It will compare the effects (good or bad) of platelet rich plasma against the effects of a placebo (normal saline) on the condition being studied in this research.

#### How long will you be in the study?

We think you will be in this study for 1 year after surgery. The total time includes 5 office visits (one pre-operative and 4 follow-up visits) over a period of 1 year after surgery. You will also participate in Occupational Therapy, as is the standard of care after surgery. Imaging (x-rays and MR Arthrogram) will take place at your pre-operative visit and at your 6-month post-operative visit. These studies are performed, no matter your treatment group, within the standard of care.

# 3. WHAT ARE THE POSSIBLE RISKS?

Risks of procedures performed solely for research purposes are described in a table attached to the end of this consent form as Appendix B. Side effects and risks of standard of care procedures are not described in this consent form.

This section describes the possible risks and/or discomforts we anticipate you could experience that are related to the study procedures. This section includes risks for patients randomized to Group B, the PRP treatment group.

Treatment with PRP uses the patient's own blood, so there is no risk of allergy/immune reaction or disease transmission. The side effects and complications of treatment with PRP are extremely rare and include pain and infection. To minimize risk of pain, treatment with PRP will occur after arthroscopic debridement while under anesthesia. The sample of blood needed for treatment (approximately 9 cc) will be withdrawn from the patient's IV during the surgery immediately prior to use. Administration will occur through the same incision used for scope placement and will therefore not require any additional incisions or injection sites.

As with any intervention, there is a small risk of infection from the site of administration. These infections (less than 1 % chance) are often treated successfully with oral antibiotics.

#### **Unknown Risks**

There may be other side effects or risks that we cannot predict. Many side effects may go away shortly after the study medication or procedure is stopped. However, in some cases they can be serious, long-lasting, permanent, and/or fatal.

#### Follow-up Visit for Discontinuing Participants

While you are free to discontinue your participation at any time, we encourage you to complete a Final Study Visit. During this visit, we will collect safety data, and discuss any information that may be important to share with your treating physician.

**Approval Date: 1/30/2019** 

# Incidental Findings

It is possible that the research procedures could uncover information related to your health that you did not know about before and that is unrelated to the Study. Some of these findings may be too preliminary to share. Cedars-Sinai will carefully consider the research findings and determine if they should be shared with you. Research findings would only be shared with you if such sharing is approved by the Cedars-Sinai IRB and is permitted by applicable law. In some cases, additional clinical testing may be required. The cost of any additional testing and any related treatment will be your responsibility.

# 4. ARE THERE BENEFITS IN TAKING PART IN THE STUDY?

If you agree to take part in this research study, there may or may not be direct medical benefit to you. The possible benefits of taking part in the research study are improved wrist function and decreased pain. However, no benefit is guaranteed. It is possible that your condition may remain unchanged or even get worse.

We hope the information learned from this research study will benefit other individuals with triangular fibrocartilage complex tears in the future by helping us to learn about treatment with platelet rich plasma after arthroscopic debridement.

#### 5. WHY WOULD MY PARTICIPATION BE STOPPED?

Your participation in this study may be stopped at any time by the researcher or the sponsor without your consent for any reason, including:

- The study is stopped or suspended;
- Funding for the study is reduced, stopped or withdrawn;
- If it is in your best interest;
- You do not consent to continue in the study after being told of changes in the research that may affect you;
- You do not follow the study procedures;
- After enrollment you have alternative treatment that would otherwise affect the study questionnaire/outcome data;
- If you do not complete scheduled follow-up visits per protocol;
- You do not undergo surgical treatment, if deemed unwarranted by the Investigator

You may choose (or you may be required) to withdraw from *certain parts* of the study, but invited to continue with other parts. For example, you might stop taking the questionnaires, but continue with follow-up visits or allow us to continue to collect data from your medical records. Separate written consent will be requested if your continued participation will involve procedures not described in this consent form.

#### 6. ARE THERE ANY OTHER OPTIONS?

Your participation is voluntary so you have the right to decline to participate or to withdraw from this research study at any time without any penalty or loss of benefits to which you would be

Approval Date: 1/30/2019

entitled outside of the study. Choosing not to participate will not affect the care you receive at Cedars-Sinai Health System.

If you decide not to take part in this study, you have other choices. For example:

- you may choose to be treated following the usual clinical approach
- you may choose to take part in a different study at CSMC or elsewhere, if one is available
- you could decide not to be treated.

The researcher will discuss these options and their risks and benefits with you.

# 7. <u>WILL MY INFORMATION BE KEPT CONFIDENTIAL?</u>

We will do our best to make sure that the personal information collected as part of this study is kept private. However, we cannot guarantee total privacy. A copy of your research consent and authorization forms may be filed in your electronic medical record at CSMC. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other identifiable personal information will not be used. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include: accrediting agencies, government and regulatory groups (such as Food and Drug Administration (FDA), Office for Human Research Protections (OHRP), etc.), safety monitors, companies that sponsor the study, and authorized representatives of the sponsor.

You will be asked to sign a separate "Authorization Form" that outlines with whom your information may be shared for the purposes of this research and under what circumstances.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

# 8. WHAT IF I BECOME ILL OR INJURED BECAUSE OF TAKING PART IN THIS STUDY?

Contact your researcher at once if you feel that you are ill or have been injured because of taking part in this study. If it is a medical emergency, call 911 or go to an emergency room. Promptly notify your researcher of your situation at the phone number listed on page 1 of this consent form.

# Who pays for my research related illness or injury?

Cedars-Sinai has no plans to pay for costs associated with the treatment of research-related injury or illness. We will make every effort to seek reimbursement from your health plan. However, you will be responsible for any deductibles and co-payments required under your health plan and for any claims ultimately denied by your health plan. Financial assistance may be available under Cedars-Sinai's Charity Care Policy and Procedure. If you feel that you have had a research-related injury and need financial assistance, please contact the IRB Office at 310-423-3783.

Approval Date: 1/30/2019

# 9. <u>FINANCIAL CONSIDERATIONS</u>

#### Costs of Participation

Please review the attached flowchart for a listing of items, drugs and services that will be billed to you and/or your insurance and those that will be covered by the study sponsor.

Standard of care procedures will be charged to you or your insurance company. You will not be charged for the use of the CASCADE Autologous Platelet System for processing of the platelet rich plasma. You remain responsible for all deductibles, co-pays, and balances under your health benefit plan.

The Researcher and/or research staff will seek pre-authorization from your insurance company for the procedures in this study. Before any study procedures are performed, pre-authorization must be received from your insurance company. If your insurance company denies coverage, you may decline to participate in the Study or you may choose to pay out of pocket. You should check with your health benefit plan if you have questions or concerns about your insurance coverage.

#### Compensation for Participating

You will not be paid for taking part in this research study.

#### Financial Interest in the Research

The PI and institution have no potential financial conflict of interest with respect to this study.

Dr. David Kulber is a board member for MTF Biologics, the makers of the CASCADE Autologous Platelet System used to process the platelet rich plasma. He has not and will not receive payment from the company for the purposes of this study.

# 10. WHAT IF I HAVE QUESTIONS OR PROBLEMS?

Please contact one of the investigators listed on the first page of this form for questions or concerns about the research.

If you have questions, problems, or concerns that you want to discuss with someone who is not associated with this study, or want to offer suggestions or feedback, please contact:

Cedars-Sinai Human Research Protection Program (HRPP) Phone: (310) 423-3783 Email: ResearchConcerns@cshs.org

The Cedars-Sinai HRPP has been established to protect the rights and welfare of research participants. You may also contact the Cedars-Sinai HRPP if you want to offer input or obtain information regarding the study.

Approval Date: 1/30/2019

# 11. CONSENT PROVISIONS

If you sign this form below, it means that:

- (1) You have taken the time to carefully read and understand the information presented in this informed consent form; you should discuss it with others, and if appropriate seek a second opinion to make an informed decision;
- (2) The information concerning the research study and its involved procedures has been fully explained to you and your questions have been answered to your satisfaction;
- (3) You have received and understand all of the information you desire regarding your participation in the research study;
- (4) You have considered the potential risks, any anticipated benefits and alternatives (and their relative risks and benefits) of participation;
- (5) You are voluntarily agreeing to participate in this research study;
- (6) You understand that by consenting to participate in the research, you are not giving up any of your legal rights;
- (7) You understand that you have the right to be informed of significant new findings related to this research study which may affect your willingness to continue participating in this study; and
- (8) You have been provided with a copy of the "Experimental Subject's Bill of Rights", if applicable to this research study, and have been provided with an opportunity to ask questions regarding the Bill of Rights.

We will give you a copy of this signed and dated consent form and a signed copy of the Experimental Subject's Bill of Rights.

| SIGNATURE BY THE PARTICIPANT: | | |
|---|---|---|
| Name of Participant (Print) | Signature of Participant | Date of Signature |
| SIGNATURE BY THE INVEST | TIGATOR: | |
| I have personally explained the resquestions, and attest that he/she fre provided with the Experimental Su | eely consents to participate. The pa | - |
| Name of Investigator (Print) | | |
| Signature of the Investigator Who | Obtained Consent | Date of Signature |

Approval Date: 1/30/2019



#### **EXPERIMENTAL SUBJECT'S BILL OF RIGHTS**

In accordance with California Health and Safety Code 24172, any person who is required to consent to participate as a subject in a research study involving a medical experiment or who is requested to consent on behalf of another has the right to:

- 1. Be informed of the nature and purpose of the experiment.
- 2. Be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized.
- 3. Be given a description of any attendant discomforts and risks to the subject reasonably to be expected from the experiment.
- 4. Be given an explanation of any benefits to the subject reasonably to be expected from the experiment, if applicable.
- 5. Be given a disclosure of any appropriate alternative procedures, drugs or devices that might be advantageous to the subject, and their relative risks and benefits.
- 6. Be informed of the avenues of medical treatment, if any, available to the subject after the experiment if complications should arise.
- 7. Be given an opportunity to ask any questions concerning the experiment or the procedure involved.
- 8. Be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation in the medical experiment without prejudice.
- 9. Be given a copy of any signed and dated written consent form used in relation to the experiment.
- 10. Be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion, or undue influence on the subject's decision.

| Signature of Experimental Subject | Date |
|-----------------------------------|------|

**Approval Date: 1/30/2019** 

# **Distribution instruction for researchers:**

The signed (i) Consent form, (ii) Authorization for Use and Disclosure of Identifiable Health Information and (iii) "Experimental Subject's Bill of Rights" (the latter required if the research study involves medical interventions) should be distributed to:

- 1) Medical Chart
- 2) Research Participant
- 3) Pharmacy
- 4) Principal Investigator's research records (original)

Approval Date: 1/30/2019

# APPENDIX A: FLOWCHART OF PROCEDURES- Medicare Coverage Analysis (MCA) Review

| FLOWCHART OF PROCEDURES | | | | | | |
|---|---|---|---|---|---|---|
| Procedures | Screening<br>Visit | Procedure | Visit #2<br>Month 1 | Visit #3<br>Month 3 | Visit #4<br>Month 6 | Visit #5<br>Year 1 |
| Informed consent | R | | | | | |
| Physical Exam | S | - | S | S | S | S |
| Demographics, Medical History | S | | S | S | S | S |
| Medical Photography | S | S | S | S | S | S |
| Randomization (during surgery) | | R | | | | |
| Platelet Rich Plasma (PRP) processed using<br>the Cascade Autologous Platelet System<br>or placebo per randomization | | R | | | | |
| Hand Imaging (X-ray) | S | | | | S | |
| MR Arthrogram | S | | | | S | |
| Surgery with athroscopy | | S | | | | |
| Two questionnaires per visit: Patient-rated Wrist Evaluation (PRWE) and Modified Mayo Wrist Score | R | | R | R | R | R |

# **LEGEND**

 $\overline{\mathbf{R}} = \text{Research item/procedure done only for research purposes and covered by the study}$ 

S = Standard of care item/procedure that is part of regular care and billed to the patient/insuranc

**Approval Date: 1/30/2019** 

# APPENDIX B: Detailed Description of Common Medical Procedures Performed for Research Purposes and Associated Risks

The procedures listed below are often performed as part of routine care for a person with your condition. They are being repeated, or performed more frequently as part of this research. However, the risks associated with each procedure should be comparable to what you would experience even if you were undergoing the procedure outside this research study.

| Study Procedure | Related Risks |
|---|---|
| Physical Exam: Includes height, weight, vital signs (heart | There are no physical risks associated with these procedures. |
| rate and blood pressure) | |
| Concomitant Medications: You will be asked about your | There are no physical risks associated with these procedures. |
| previous and current medications that you take. | |
| Medical History Review: You will be asked about your | There are no physical risks associated with this procedure. |
| medical and surgical history with attention to smoking and | |
| alcohol habits, and your physical activity | |
| Questionnaires: You will be asked to complete two | If you feel uncomfortable or embarrassed answering any question, |
| questionnaires at visit. We will ask you questions to | you may skip it. The questionnaire will contain your research |
| evaluate pain and function after surgery. We think it | identification number. |
| should take about 15 minutes to complete the | |
| questionnaires. One questionnaire will be self- | |
| administered. The other questionnaire will be completed | |
| with the help of a study team member in a face-to-face | |
| interview. | |
| Demographic Information: You will be asked about | There are no physical risks associated with these procedures |
| your age, gender, race, ethnicity | |